CLINICAL TRIAL: NCT02596152
Title: Comparison of 12-week Mini-trampoline Intervention With a Nordic Walking Intervention: Balance, Fitness and Neuropsychological Effects
Brief Title: Mini-trampoline Intervention vs. Nordic Walking: Balance, Fitness and Neuropsychological Effects
Acronym: TraWaFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arno Schmidt-Trucksäss (Other)
Responsible Party: Sponsor-Investigator, Arno Schmidt-Trucksäss, Prof. Dr. Arno Schmidt-Trucksäss, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EKNZ 2015-231/232
Record Dates: First submitted 2015-10-30; First posted 2015-11-04 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Overweight; Obesity
Keywords: balance; strength; barriers towards exercise; quality of life; body dissatisfaction; executive functions; eating behavior; fitness
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior | interventions — Nordic Walking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mini-trampoline (Experimental): participants allocated to this group will participate in a 12-week mini-trampoline group instructed training twice a week.
  Interventions: Other: mini-trampoline
- Nordic Walking (Active Comparator): participants allocated to this group will participate in a 12-week Nordic Walking group instructed training twice a week.
  Interventions: Other: Nordic Walking

INTERVENTIONS:
Other: mini-trampoline — Intervention period lasts 12 weeks, training is group instructed, twice weekly. Training sessions are one hour each. The training intensity of the two interventional arms is comparable. The training progression is defined in advance.
  Arms: Mini-trampoline
Other: Nordic Walking — Intervention period lasts 12 weeks, training is group instructed, twice weekly. Training sessions are one hour each. The training intensity of the two interventional arms is comparable. The training progression is defined in advance.
  Arms: Nordic Walking

SUMMARY:
The effects of mini-trampoline training on balance, cardiorespiratory fitness, strength and neuropsychological parameters in an overweight or obese population are unknown. The aim of this 2-arm randomized controlled trial is to compare the effects of a 12-week mini-trampoline training and a 12-week nordic walking training on balance, fitness and strength in overweight/obese individuals.

DETAILED DESCRIPTION:
A growing body of literature suggests, that obesity is not only associated with medical conditions such as diabetes, but also linked to altered gait, impaired balance and a greater likelihood of falls. Weight reduction has been shown to improve balance controle. Methods to increase physical activity are largely not accepted in this population and those which conserve the musculoskeletal system are rare. Physical activity has been shown to influence mood, quality of life and eating behavior. Mini-trampoline training has been shown to enhance stability and increase fitness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Body Mass Index ≥25 kg/m2
* ≤ 1h regular exercise/ physical activity per week

Exclusion Criteria:

* cardiovascular or other chronic diseases not permitting sports participation
* inability to follow the procedures of the study (e.g. due to dementia)
* neurological disorders limiting balance or medications impairing balance
* hypertensive blood pressure not permitting exercise (>180/100 mmHg)
* medication: beta-blocking agents which reduce cardiac adaption abilities to exercise
* known pregnancy with contraindications for exercise according to the guidelines of the American College of Obstetricians and Gynecologists

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Postural sway | assessed twice: before and after the intervention (12 weeks)
  COPspeed (Center of pressure speed measured on a force plate in cm/sec) measured on a force plate in quiet stance with eyes closed

SECONDARY OUTCOMES:
peak oxygen uptake | assessed twice: before and after the intervention (12 weeks)
  (VO2 peak in ml/kg/min)
submaximal heart rate at 50 Watts | assessed twice: before and after the intervention (12 weeks)
  (HR at 50 Watts in beats/min)
maximal work | assessed twice: before and after the intervention (12 weeks)
  (Watts on bicycle ergometer)
dynamic core strength | assessed twice: before and after the intervention (12 weeks)
  (Nm/kg on dynamometer)
lower body explosive strength | assessed twice: before and after the intervention (12 weeks)
  (seconds on chair rise test)
lower body functional endurance | assessed twice: before and after the intervention (12 weeks)
  (repetitions during 30-second-chair rise test)
isokinetic plantar flexion strength | assessed twice: before and after the intervention (12 weeks)
  (Nm/kg on dynamometer)
functional balance | assessed twice: before and after the intervention (12 weeks)
  (cm in reach test)
body fat mass | assessed twice: before and after the intervention (12 weeks)
  (in kg)
waist circumference | assessed twice: before and after the intervention (12 weeks)
  (in cm)
motivation and barriers | assessed twice: before and after the intervention (12 weeks)
  (score on questionnaire)
mood | assessed twice: before and after the intervention (12 weeks)
  (score on multidimensional mood questionnaire)
weight adjusted quality of life | assessed twice: before and after the intervention (12 weeks)
  (score on IWQOL questionnaire)
body dissatisfaction | assessed twice: before and after the intervention (12 weeks)
  (score on Figure Rating Scale)
eating behavior | assessed twice: before and after the intervention (12 weeks)
  (score on FEV questionnaire)
attention | assessed twice: before and after the intervention (12 weeks)
  (score on the digit span test)
cognitive flexibility | assessed twice: before and after the intervention (12 weeks)
  (seconds during the Trail making test)
executive planning function | assessed twice: before and after the intervention (12 weeks)
  (score in the Tower of London Test (computer based version))
behavioral shift and inhibition | assessed twice: before and after the intervention (12 weeks)
  (number of mistakes in the Inhib Test (computer based version))
body muscle mass | assessed twice: before and after the intervention (12 weeks)
  (in kg)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Department of Sport, Exercise and Health, Basel, Switzerland